CLINICAL TRIAL: NCT02123719
Title: Outcomes Analysis of Laparoscopic Incisional Hernia Repair and Risk Factors for Hernia Recurrence in Liver Transplant Patients
Brief Title: Laparoscopic Incisional Hernia Repair in Liver Transplant Patients
Status: Completed | Type: Observational
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Matthias Biebl, Priv.-Doz. M.D., Medical University Innsbruck
Other Study IDs: 1304197302
Record Dates: First submitted 2014-04-24; First posted 2014-04-25 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-04

CONDITIONS: Hernia Recurrence Post Laparoscopic Incisional Hernia Repair in Liver Transplant Versus Non-transplant Patients.
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients post liver transplantation: Patients after liver transplantation
  Interventions: Other: Surgery
- Control group: Patients with an abdominal incisional hernia without a history of immunosuppresion
  Interventions: Other: Surgery

INTERVENTIONS:
Other: Surgery

SUMMARY:
Retrospective analysis of patients undergoing laparoscopic incisional hernia repair.

Study group: Patients with incisional hernia post liver transplantation Control group: Patients with incisional hernia post any other laparotomy in the upper quadrant.

Primary study outcome parameter: Risk of hernia recurrence. Secondary study outcome parameters: - Hernia repair-related infection rate

- Postoperative morbidity Statistical analysis: Comparison of study versus control group, univariate and multivariate analysis, Chi² and Mann-Whitney-U tests. P-values <0.05 were considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Incisional hernia
* Laparoscopic repair possible

Exclusion Criteria:

* Other types of ventral hernias
* Laparoscopy not possible

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with incisional hernia post liver transplantation
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Hernia recurrence post laparoscopic incisional hernia repair | 1 - 74 months post surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Innsbruck, Innsbruck, Tyrol, Austria